CLINICAL TRIAL: NCT05147935
Title: Adding Specialist Palliative Care to Transplantation Pilot Trial
Acronym: ASPECT-Pilot
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Myrick C. Shinall, Jr., MD, PhD, Study Principal Investigator Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ASPECT-Pilot
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: End Stage Liver DIsease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Specialist Palliative Care (Experimental): All patients will be assigned to receive the intervention, consisting of two outpatient palliative care visits at Vanderbilt University Medical Center (VUMC).
  Interventions: Behavioral: Palliative Care Consultation

INTERVENTIONS:
Behavioral: Palliative Care Consultation — In person or telehealth clinic visit with palliative care physician or nurse practitioner

SUMMARY:
Specialist palliative care has been shown to be beneficial for patients experiencing serious illness, but has not been studied for patients being evaluated for liver transplantation. The investigators hope in the future to design a multi-center trial of a specialist palliative care intervention to measure the effects of specialist palliative care for patients undergoing liver transplant evaluation. This project represents a pilot to gather needed information to design such a future study.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 18 years or greater) undergoing evaluation for liver transplantation at Vanderbilt University Medical Center

Exclusion Criteria:

1. Patient does not speak English fluently
2. Patient lacks a telephone
3. Patient is a prisoner
4. Patient is deaf
5. Patient currently receives specialist palliative care
6. Patient is not a resident of Tennessee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention | 2 months
  Score on the Acceptability of Intervention Measure (AIM) which measures how acceptable participants find the intervention with 4 questions, each scored 1-5 with higher scores indicating greater acceptability.
Appropriateness of Intervention | 2 months
  Score on the Intervention Appropriateness Measure (IAM), which measures how appropriate the palliative care intervention seems to the study participants with 4 questions, each scored 1-5 with higher scores indicating higher appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Myrick C Shinall, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No